CLINICAL TRIAL: NCT02100748
Title: A Phase 2, Multicenter, Randomized, Double-blind, Multiple-dose, Adaptive, Placebo- and Active-controlled Study of TRV130 for the Treatment of Acute Postoperative Pain After Bunionectomy
Brief Title: A Study of TRV130 for the Treatment of Pain After Bunionectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trevena Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CP130-2001
Record Dates: First submitted 2014-03-23; First posted 2014-04-01 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Acute Pain
Keywords: moderate to severe acute pain; bunionectomy
MeSH Terms: conditions — Acute Pain | interventions — ((3-methoxythiophen-2-yl)methyl)((2-(9-(pyridin-2-yl)-6-oxaspiro(4.5)decan-9-yl)ethyl))amine; Morphine; Glucose; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- TRV130 1 mg (Experimental): TRV130 1 mg IV Q4H x 48 h
  Interventions: Drug: TRV130
- TRV130 2 mg (Experimental): TRV130 2 mg IV Q4H x 48 h
  Interventions: Drug: TRV130
- TRV130 3 mg (Experimental): TRV130 3 mg IV Q4H x 48 h
  Interventions: Drug: TRV130
- TRV130 4 mg (Experimental): TRV130 4 mg IV Q4H x 48 h
  Interventions: Drug: TRV130
- Morphine (Active Comparator): Morphine 4 mg IV Q4H x 48 h
  Interventions: Drug: Morphine
- Placebo (Placebo Comparator): Placebo (D5W) IV Q4H x 48 h
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRV130 — TRV130 1 - 4 mg will be administered every 4 hours
  Arms: TRV130 1 mg; TRV130 2 mg; TRV130 3 mg; TRV130 4 mg
Drug: Morphine — Morphine 4 mg will be administered every 4 hours
  Other Names: Morphine sulphate
  Arms: Morphine
Drug: Placebo — Placebo will be administered every 4 hours
  Other Names: Dextrose 5% in water; D5W
  Arms: Placebo

SUMMARY:
The primary objective is to evaluate the analgesic efficacy of IV TRV130 compared with placebo in patients with acute postoperative pain after bunionectomy.

DETAILED DESCRIPTION:
The primary objective is to evaluate the analgesic efficacy of IV TRV130 compared with placebo in patients with acute postoperative pain after bunionectomy. The results section also includes data from the morphine arms.

ELIGIBILITY:
Inclusion Criteria:

* Has undergone primary, unilateral, first metatarsal bunionectomy (osteotomy and internal fixation) with no additional collateral procedures.
* Experiences a pain intensity rating of ≥ 4 on an 11 point NRS
* Able to provide written informed consent before any study procedure.

Exclusion Criteria:

* ASA Physical Status Classification System classification of P3 or worse
* Has surgical or post-surgical complications.
* Has clinically significant medical conditions or history of such conditions that may interfere with the interpretation of efficacy, safety, or tolerability data obtained in the trial, or may interfere with the absorption, distribution, metabolism, or excretion of drugs.
* Has previously participated in another TRV130 clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franck Skobieranda, MD, Study Director — Trevena Inc.
Locations (4):
- United States (4):
  - Premier Research, Phoenix, Arizona
  - Chesapeake Research Group, Pasadena, Maryland
  - Premier Research, Austin, Texas
  - Jean Brown Research, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A - TRV130 1 mg: TRV130 1 mg IV Q4H x 48 h
  TRV130: TRV130 1 - 4 mg will be administered every 4 hours
- Part A - TRV130 2 mg: TRV130 2 mg IV Q4H x 48 h
  TRV130: TRV130 1 - 4 mg will be administered every 4 hours
- Part A - TRV130 3 mg: TRV130 3 mg IV Q4H x 48 h
  TRV130: TRV130 1 - 4 mg will be administered every 4 hours
- Part A - TRV130 4 mg: TRV130 4 mg IV Q4H x 48 h
  TRV130: TRV130 1 - 4 mg will be administered every 4 hours
- Part A - Morphine; Part B - Morphine: Morphine 4 mg IV Q4H x 48 h
  Morphine: Morphine 4 mg will be administered every 4 hours
- Part A - Placebo: Placebo (D5W) IV Q4H x 48 h
  Placebo: Placebo will be administered every 4 hours
- Part B - TRV130 0.5 mg: TRV130 0.5 mg IV Q3H x 48 h
  TRV130: TRV130 0.5 - 4 mg will be administered every 3 hours
- Part B - TRV130 1 mg: TRV130 1 mg IV Q3H x 48 h
  TRV130: TRV130 0.5 - 4 mg will be administered every 3 hours
- Part B - TRV130 2 mg: TRV130 2 mg IV Q3H x 48 h
  TRV130: TRV130 0.5 - 4 mg will be administered every 3 hours
- Part B - TRV130 3 mg: TRV130 3 mg IV Q3H x 48 h
  TRV130: TRV130 0.5 - 4 mg will be administered every 3 hours
- Part B - Placebo: Placebo (D5W) IV Q3H x 48 h
  Placebo: Placebo will be administered every 3 hours
Period: Overall Study
Arm/Group | Part A - TRV130 1 mg | Part A - TRV130 2 mg | Part A - TRV130 3 mg | Part A - TRV130 4 mg | Part A - Morphine | Part A - Placebo | Part B - TRV130 0.5 mg | Part B - TRV130 1 mg | Part B - TRV130 2 mg | Part B - TRV130 3 mg | Part B - Placebo | Part B - Morphine
Started | 25 | 24 | 22 | 22 | 25 | 23 | 20 | 38 | 36 | 31 | 28 | 39
Completed | 23 | 23 | 21 | 21 | 23 | 23 | 18 | 34 | 33 | 29 | 26 | 39
Not Completed | 2 | 1 | 1 | 1 | 2 | 0 | 2 | 4 | 3 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A - TRV130 1 mg | Part A - TRV130 2 mg | Part A - TRV130 3 mg | Part A - TRV130 4 mg | Part A - Morphine | Part A - Placebo | Part B - TRV130 0.5 mg | Part B - TRV130 1 mg | Part B - TRV130 2 mg | Part B - TRV130 3 mg | Part B - Placebo | Part B - Morphine | Total
Number analyzed (Participants) | 25 | 24 | 22 | 22 | 25 | 23 | 20 | 38 | 36 | 31 | 28 | 39 | 333
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (12.52) | 41.8 (12.06) | 40.3 (13.33) | 42.1 (13.66) | 41.5 (12.53) | 43.5 (9.94) | 38.6 (11.38) | 43.3 (11.02) | 36.7 (12.23) | 37.5 (10.58) | 39.9 (11.04) | 42.6 (13.09) | 41.2 (12.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 19 | 20 | 24 | 21 | 18 | 34 | 32 | 29 | 25 | 31 | 297
  Male | 3 | 2 | 3 | 2 | 1 | 2 | 2 | 4 | 4 | 2 | 3 | 8 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 22 | 22 | 16 | 21 | 22 | 17 | 16 | 28 | 24 | 24 | 22 | 27 | 261
  Black | 3 | 2 | 5 | 0 | 3 | 6 | 2 | 6 | 10 | 5 | 5 | 11 | 58
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 5
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 4
  Other - Race | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 5
  Hispanic or Latino | 9 | 8 | 3 | 7 | 10 | 6 | 3 | 8 | 8 | 11 | 6 | 9 | 88
  Not Hispanic or Latino | 16 | 16 | 19 | 15 | 15 | 17 | 17 | 30 | 28 | 20 | 22 | 30 | 245
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 22 | 22 | 25 | 23 | 20 | 38 | 36 | 31 | 28 | 39 | 333

OUTCOME MEASURES:

1. Primary Outcome: Time Weighted Average (TWA) Change From Baseline in Pain Score Over 48 Hours Between TRV130 and Placebo
Description: Pain intensity will be evaluated using an 11-point (0-10) Numeric Pain Rating Scale (NPRS), with higher numbers indicating a higher pain intensity, administered over 48 hours. Time weighted average change from baseline is calculated using the following: time weighted sum of pain intensity differences (SPID) divided by a constant (48 hours) to yield values on the 0-10 NPRS.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A - TRV130 1 mg | Part A - TRV130 2 mg | Part A - TRV130 3 mg | Part A - TRV130 4 mg | Part A - Morphine | Part A - Placebo | Part B - TRV130 0.5 mg | Part B - TRV130 1 mg | Part B - TRV130 2 mg | Part B - TRV130 3 mg | Part B - Placebo | Part B - Morphine
Number analyzed (Participants) | 25 | 24 | 22 | 22 | 25 | 23 | 20 | 38 | 36 | 31 | 28 | 39
score on a scale | -3.1 (2.11) | -3.1 (2.25) | -2.6 (1.82) | -3.3 (1.51) | -4.1 (2.02) | -3.2 (1.79) | -3.0 (2.36) | -2.9 (2.64) | -3.7 (2.10) | -5.0 (2.14) | -2.8 (2.12) | -4.0 (1.89)

ADVERSE EVENTS:
Arm/Group | Part A - TRV130 1 mg | Part A - TRV130 2 mg | Part A - TRV130 3 mg | Part A - TRV130 4 mg | Part A - Morphine | Part A - Placebo | Part B - TRV130 0.5 mg | Part B - TRV130 1 mg | Part B - TRV130 2 mg | Part B - TRV130 3 mg | Part B - Placebo | Part B - Morphine
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24 | 0/22 | 0/22 | 0/25 | 0/23 | 0/20 | 0/38 | 0/36 | 0/31 | 0/28 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24 | 0/22 | 0/22 | 0/25 | 0/23 | 0/20 | 0/38 | 0/36 | 0/31 | 0/28 | 0/39
Other Adverse Events (participants affected / at risk) | 22/25 | 21/24 | 20/22 | 22/22 | 23/25 | 11/23 | 16/20 | 31/38 | 31/36 | 28/31 | 20/28 | 31/39
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A - TRV130 1 mg (N=25) | Part A - TRV130 2 mg (N=24) | Part A - TRV130 3 mg (N=22) | Part A - TRV130 4 mg (N=22) | Part A - Morphine (N=25) | Part A - Placebo (N=23) | Part B - TRV130 0.5 mg (N=20) | Part B - TRV130 1 mg (N=38) | Part B - TRV130 2 mg (N=36) | Part B - TRV130 3 mg (N=31) | Part B - Placebo (N=28) | Part B - Morphine (N=39)
Nausea (Gastrointestinal disorders) | 9 | 14 | 11 | 16 | 16 | 3 | 7 | 13 | 20 | 23 | 7 | 22
Dizziness (Nervous system disorders) | 9 | 13 | 13 | 17 | 11 | 2 | 4 | 22 | 17 | 18 | 4 | 17
Vomiting (Gastrointestinal disorders) | 2 | 5 | 7 | 11 | 11 | 1 | 0 | 4 | 10 | 17 | 0 | 12
Headache (Nervous system disorders) | 5 | 6 | 4 | 5 | 7 | 3 | 5 | 10 | 7 | 7 | 5 | 9
Somnolence (Nervous system disorders) | 4 | 2 | 9 | 4 | 8 | 1 | 4 | 5 | 4 | 4 | 3 | 7
Constipation (Gastrointestinal disorders) | 3 | 2 | 2 | 4 | 4 | 1 | 2 | 6 | 3 | 5 | 1 | 2
Hot Flash (Vascular disorders) | 2 | 3 | 3 | 6 | 0 | 0 | 0 | 2 | 5 | 4 | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 3 | 4 | 1 | 0 | 1 | 4 | 3 | 2 | 2
Dry Mouth (Gastrointestinal disorders) | 1 | 3 | 2 | 1 | 2 | 0 | 0 | 2 | 4 | 1 | 2 | 1
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 4 | 1 | 0 | 0 | 0 | 3 | 5 | 0 | 1
Flushing (Vascular disorders) | 1 | 3 | 1 | 1 | 0 | 0 | 0 | 3 | 6 | 3 | 0 | 4
Paraesthesia (Nervous system disorders) | 0 | 3 | 1 | 2 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0 | 1 | 0 | 1 | 0 | 2 | 2 | 1 | 2
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Feeling Hot (General disorders) | 0 | 0 | 2 | 4 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus Generalized (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 4 | 0 | 1 | 1 | 1 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other